CLINICAL TRIAL: NCT06844370
Title: Home Initiation and Monitoring of Non-invasive Ventilation (NIV) Versus Hospital-based Care in People with Motor Neurone Disease (MND) : a Randomised Control Trial (RCT) and Qualitative Study
Brief Title: Home Versus Hospital Based NIV Care in MND
Acronym: HoHoNIV
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Papworth Hospital NHS Foundation Trust (Other Government)
Collaborators: University of Nottingham (Other); MND Association (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: P03084
Record Dates: First submitted 2024-03-14; First posted 2025-02-25 (Actual); Last update posted 2025-02-25 (Actual); Status verified 2025-02

CONDITIONS: Motor Neurone Disease; Respiratory Insufficiency
Keywords: non invasive ventilation
MeSH Terms: conditions — Amyotrophic Lateral Sclerosis; Respiratory Insufficiency | interventions — Noninvasive Ventilation

STUDY DESIGN:
Intervention Model Description: Random allocation to either home or hospital based treatment
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Home initiation of NIV (Other): Initiation of NIV at home and follow up by home visits and telemonitoring
  Interventions: Other: Non-invasive ventilation
- Hospital initiation of NIV (Other): Initiation of NIV at hospital with monitoring at outpatient visits
  Interventions: Other: Non-invasive ventilation

INTERVENTIONS:
Other: Non-invasive ventilation — Providing ventilation support through non-invasive means

SUMMARY:
Non-invasive ventilation (NIV) is commonly offered to people with Motor Neurone Disease (MND) who have breathing difficulties. It improves their quality of life and can prolong life by 6 months or more. It is initially used at night and typically set up during a hospital admission. By the time that they develop respiratory failure and need to start NIV, however, most patients require wheelchairs or have other significant health problems. Repeated travel to hospitals is increasingly difficult with increasing disability. It is possible to start and monitor NIV treatment at home. This may be more convenient for selected patients, though starting NIV is quite complex; it is not known if home treatment is as safe and effective as hospital-based treatment.

To establish this, 60 patients with MND who have indications for NIV will be recruited. They will be randomly allocated to a home-based treatment (home NIV set up plus home visits supported by telemonitoring) or hospital-based care (inpatient NIV set up plus outpatient NIV monitoring) and followed up at 1, 4 and 7 months. Alongside measures of treatment effectiveness, assessment of patient and carer preferences, quality of life, and cost-effectiveness will be undertaken.

In the additional qualitative part on this study, interviews with patients who took part in the main study and their carers will be conducted to understand in more depth their perspective on what makes for a good or bad experience with NIV, how the environment (home vs hospital) influences their NIV experience and what personal factors determine NIV use. Findings from the interviews will inform the design of a truly patient-centred NIV service.

ELIGIBILITY:
Inclusion Criteria:

* Adults with a diagnosis of Motor Neurone Disease confirmed by a neurologist specialising in MND.
* Indications to NIV: daytime pCO2 >6.0 kPa or/and symptoms of ventilatory failure (e.g. orthopnoea, paroxysmal nocturnal dyspnoea, morning drowsiness) in the presence of significant diaphragmatic weakness confirmed by respiratory muscle tests

Exclusion Criteria:

* Cognitive impairment precluding understanding of the study protocol and valid consent
* Severe co-morbidities (e.g. decompensated heart failure, severe chronic obstructive pulmonary disease (COPD), morbid obesity) causing or contributing to respiratory failure
* Immediate need to start NIV (<24hrs) and/or acute illness requiring inpatient treatment e.g. intravenous antibiotics for pneumonia (in addition to the need for NIV)
* Lack of a sufficient social/professional network to support NIV application at home
* Not wishing to accept home NIV

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2024-03-06 (Actual); Primary Completion 2026-02 (Estimated); Study Completion 2026-09 (Estimated)

PRIMARY OUTCOMES:
Control of respiratory failure defined by daytime partial pressure of carbon dioxide (PaCO2) | measured at 1,4,7 months following NIV initiation
  Daytime PaCO2 measured by arterial puncture
Patients and carers experiences of starting and managing NIV, and factors that relate to NIV concordance and acceptance. | measured at 4 weeks since starting NIV
  Semi-structured interview with patients and their carers

SECONDARY OUTCOMES:
NIV acceptance | 1 month
  Percent of patients using NIV for >=4hrs/night
NIV concordance | 1 , 4 and 7 months
  NIV adherence (machine usage in hours/24hours)
Survival | Survival since NIV initiation
  Survival (in months)
Admissions | Up to 7 months from initiation of NIV
  Number of additional planned and emergency hospital admissions
NIV setting changes | 1 , 4 and 7 months
  Number of NIV setting changes required
Cost effectiveness | Up to 7 months from initiation of NIV
  Absolute costs and costs in relation to quality-adjusted life-years (using EQ-5D)
Nocturnal oximetry | 1,4,7 months
  time spent with oxygen saturation <90%(TST90)
Other blood gas analysis measurements of hypoventilation | 1,4,7 months
  Bicarbonate
Quality of life assessment (EQ-5D-5L) | 1,4,7 ,months
  Measurement of quality of life using EQ-5D-5L questionnaire
Quality of life (SRI) | 1,4, 7 months
  Quality of life measured using Severe Respiratory Insufficiency (SRI) questionnaire
Quality of sleep | 1,4,7 ,months
  Sleep quality measured with Pittsburgh Sleep Quality Index (PSQI)
Satisfaction with NIV and healthcare interactions | 7 months
  Satisfaction with NIV and healthcare interactions measured with a visual analogue scale

CONTACTS AND LOCATIONS:
Overall Officials: Dariusz Wozniak, Principal Investigator — Royal Papworth Hospital NHS Foundation Trust
Locations (1):
- Royal Paworth Hospital, Cambridge, United Kingdom

IPD SHARING:
Plan to Share IPD: No